CLINICAL TRIAL: NCT02830412
Title: A Prospective Randomized Evaluation of an Intraoperative Electronic Reminder Module to Enhance Postoperative Nausea and Vomiting Prophylaxis Guideline Adherence
Brief Title: Intraoperative Electronic Reminder Module to Enhance Postoperative Nausea and Vomiting Prophylaxis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-1193
Record Dates: First submitted 2015-10-05; First posted 2016-07-12 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PONV Reminder (Experimental): After patient has non-cardiac surgery, the subject will have Post-Operative Nausea and Vomiting Reminder display
  Interventions: Other: Postoperative nausea and vomiting (PONV) reminder
- No PONV Reminder (No Intervention): After patient has non-cardiac surgery, the subject will not have Post-Operative Nausea and Vomiting Reminder display

INTERVENTIONS:
Other: Postoperative nausea and vomiting (PONV) reminder — The postoperative nausea and vomiting (PONV) electronic reminder will be programmed to assess the patient risk for PONV according to the risk factors identified by Apfel and Koivuranta. The PONV risk assessment and current guidelines will be displayed electronically for patients randomized to receive the reminder.
  Arms: PONV Reminder

SUMMARY:
This project intends to develop and implement an electronic reminder for post-operative nausea and vomiting (PONV) prophylaxis into the Anesthesia Record Keeping System.

Each patient will have his or her PONV risk classified based on the following risk factors: Female gender, History of PONV, History of Motion Sickness, Non-smoker and Duration of procedure > 60 minutes.

Patients will be randomized to either receive the PONV reminder or not. Those receiving the PONV reminder will have the PONV risk assessment and current guideline information for PONV prophylaxis displayed on the Anesthesia Record Keeping System (ARKS) screen at the beginning of the case.

At the end of the procedure (specific at documentation of emergence), the reminder will assess the current status of PONV prophylaxis as per anti-emetic medications administered and compare the current status to the recommended status based on published guidelines.

If the current status is compatible or exceeds the recommended status the reminder will silently document compliance.

If published guidelines suggest additional PONV prophylaxis based on the patients risk profile and a comparison with the currently documented status, an electronic reminder will appear on the ARKS screen to alert the anesthesia provider of an opportunity to enhance guideline adherence.

The reminder will not recommend a specific medication, intervention or therapy.

It will be completely the decision of the anesthesia provider if and how to modify the PONV prophylaxis for the patient.

Subjects randomized to not receive the electronic display will have it deactivated.

DETAILED DESCRIPTION:
Each patient will have his or her PONV risk classified based on the following risk factors Female gender, History of PONV or Motion Sickness, Non-smoker and Duration of procedure > 60 min utilizing information already entered into the Anesthesia Record Keeping System. Patients having 0-1 risks factors present will be low risk. 2 risks factors present are medium risk and more than 2 risk factors present are high risk.

Patients will be randomized to either receive the PONV reminder or not. Those receiving the PONV reminder will have the PONV risk assessment and current guideline information for PONV prophylaxis will be displayed on the ARKS screen at the beginning of the case.

In a second step at the end of the procedure (specific at documentation of emergence), the reminder will assess the current status of PONV prophylaxis as per anti-emetic medications administered and compare the current status to the recommended status based on published guidelines.

If the current status is compatible or exceeds the recommended status the reminder will silently document compliance.

If published guidelines suggest additional PONV prophylaxis based on the patients risk profile and a comparison with the currently documented status, an electronic reminder will appear on the ARKS screen to alert the anesthesia provider of an opportunity to enhance guideline adherence.

The reminder will display the PONV risk assessment information, current status of PONV prophylaxis as well as the information that current guidelines recommend additional PONV prophylaxis.

The reminder will not recommend a specific medication, intervention or therapy.

It will be completely the decision of the anesthesia provider if and how to modify the PONV prophylaxis for the patient.

Subjects randomized to not receive the electronic display will have it deactivated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Procedure with General Anesthesia

Exclusion Criteria:

* Postoperative admission to the Intensive Care Unit
* Postoperative fast-track to Phase II
* Patient remains sedated/intubated at the end of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | 6 hours
  Incidence of postoperative nausea and vomiting in the recovery room

SECONDARY OUTCOMES:
Duration of postoperative anesthesia care unit (PACU) stay | 6 hours
  Time to postoperative anesthesia care unit (PACU) discharge alive (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Saager leif, M.D., Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No